CLINICAL TRIAL: NCT00949429
Title: Quality of Postoperative Pain Management in Cardiac Surgical Patients
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Kasana Raksamani, Faculty of Medicine, Siriraj Hospital
Other Study IDs: Si306/2009
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; cardiac surgery; risk factors
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine the incidence and risk factors of moderate to severe pain after cardiac surgery, and compare the preoperative pain expectation and postoperative pain experience in the same patient.

DETAILED DESCRIPTION:
Objectives

1. To study the incidence of moderate to severe pain in cardiac surgical patients 48 hour postoperatively.
2. To study the risk factors of moderate to severe postoperative pain in cardiac surgical patients.
3. To compare the preoperative pain expectation and postoperative pain experience in the same patient.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for cardiac surgery in Siriraj Hospital
* age > 18

Exclusion Criteria:

* unable to communicate with the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for cardiac surgery in Siriraj Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Number of the patients having pain score more than 4 out of 10 in 48 hour postoperatively | 48 hours

SECONDARY OUTCOMES:
Risk factors of postoperative pain in cardiac surgical patients | 48 hours
Patient's preoperative pain expectation and postoperative pain experience | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kasana Raksamani, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkok, Bangkok, Thailand